CLINICAL TRIAL: NCT04512534
Title: A Phase II Study of Anti-Programmed Death-1(PD-1) Antibody Sintilimab Plus Histone Deacetylase(HDAC) Inhibitor Chidamide in Patients With Relapsed/ Refractory Peripheral T-cell Lymphoma
Brief Title: Sintilimab Combined With Chidamide in Treating Peripheral T Cell Lymphoma
Acronym: Sincerely20
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ji Dongmei, Associate Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sincerely2020
Record Dates: First submitted 2020-08-10; First posted 2020-08-13 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: relapsed/refractory peripheral T-cell lymphoma; PD-1 antibody; HDAC inhibitor; objective response rate; safety profile
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — sintilimab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Intervention Model Description: Simon's optimal two-stage design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sinitilimab+Chidamide (Experimental): Anti-PD-1 antibody Sintilimab 200mg intravenously every 3 weeks; HDAC inhibitor Chidamide 30mg orally twice every week
  Interventions: Drug: PD-1 antibody+ HDAC inhibitor

INTERVENTIONS:
Drug: PD-1 antibody+ HDAC inhibitor — Patients receive anti-PD-1 antibody Sintilimab+ HDAC inhibitor Chidamide three weeks for a cycle, detailed as follows:
  * Anti-PD-1 antibody (Sintilimab): Fixed dose of 200 mg every 3 weeks, intravenous drip (without pretreatment), infusion time: 30 minutes (no less than 20 mins, no more than 60 mins), the maximum treatment period is 2 years (up to 35 doses), complete remission（CR）patients confirmed by imaging assessment can be considered off anti-PD-1 treatment after 12 treatment cycles.
  * Chidamide: Chidamide is administered orally at a dose of 30mg (initial dose). It is recommended to be administered within 0.5h after a meal with a fixed time. Chidamide will be given until disease progression or intolerant toxicity. The maximum treatment is 2 years. If chidamide therapy requires to be continued over 2 years due to clinical benefit, the prescription/decision should be made after discussion with the principal investigator.
  Other Names: Sintilimab; Chidamide

SUMMARY:
This is a single-center, single-arm, phase 2 study to evaluate the efficacy and safety of Anti-PD-1 antibody(Sintilimab) plus HDAC inhibitor(Chidamide) in patients with relapsed/refractory peripheral T-cell lymphoma (r/r PTCL).

DETAILED DESCRIPTION:
Peripheral T-cell lymphoma accounts for 12-15% of non-Hodgkin's lymphomas in western countries, however, this number is up to 35% or more in some Asian countries, including China. According to the 2016 World Health Organization annual classification, there are 29 subtypes of peripheral T cell lymphoma, among which the most common types are peripheral T cell lymphoma non-specific type (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL) and anaplastic large cell lymphoma (ALCL). For r/r PTCL, the prognosis was poor with objective response rate range from 8-50% and median progression free survival（PFS）range from 3.2-5 months for chemotherapy. Thus, the treatment of this patient population remained clinically unmet need.

This clinical trial will be conducted under Simon's optimal two-stage design. The first stage needs 15 participants, if ≥5 participants acquire remission, the study will move on to the second stage and enroll another 36 patients to achieve a total number of 51 participants enrolled. Drop rate is assumed to be 10%, to insure 47 participants involving the efficacy evaluation statistically.

Participants will receive anti-PD-1 antibody plus HDAC inhibitor every three weeks for a cycle, until disease progression or severe/ intolerant toxicity, the maximum treatment period is 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 75 years;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
3. Pathologically confirmed relapsed/refractory Peripheral T-cell lymphoma (Including PTCL-NOS, AITL, anaplastic large cell lymphoma（ALTL）, excluding Nature Killer（NK）/T cell lymphoma);
4. At least one two-dimensional measurable lesion with a length diameter of at least 1.5cm and vertical diameter of at least 1.0cm (measured by CT or MRI);
5. Adequate medullary hematopoiesis function ( WBC≥3.5×109/L, ANC≥1.5×109/L, PLT≥80×109/L, HB≥90g/L. If the peripheral blood indicators demonstrate abnormal due to bone marrow or spleen invasion by lymphoma, Enrollment decision can be determined by the investigator as appropriate;
6. Adequate hepatic function (total serum bilirubin, ALT and AST≤1.5 times of upper limit of normal);
7. Adequate renal function (serum creatinine≤1.5 times the upper limit of normal, creatinine clearence≥50ml/min);
8. Echocardiography or radionuclide cardia functional test, LVEF≥50%;
9. Patients of child-bearing period agree to use appropriate contraception. The serum pregnancy test of women in childbearing period was negative within 2 weeks before enrollment.
10. Willingness to provide pathological tissue specimens (20 pieces of wax or paraffin tissue sections);
11. Expectation survival time over 3 months;
12. Willingness to provide written informed consent.

Exclusion Criteria:

1. Patients allergic of any drug in this regimen;
2. Previous treatment with anti-PD-1 antibody combined with HDAC inhibitor (Patients only received single agent of treatment regime or sequentially received anti-PD-1 and HDAC inhibitor are allowed to enroll);
3. Patients with clinically significant heart disease, including severe cardiac insufficiency: New York Heart Disease Association (NYHA) grade IV cardiac insufficiency, unstable angina. And myocardial infarction, congestive heart failure, and QTC interphase > 500ms which occurred before 6 month of screening;
4. Patients who have received grade II or above surgery within 3 weeks before enrollment;
5. History of other malignancy within the past 5 years (except for 1. basal cell carcinoma of the skin and 2. carcinoma in situ of the cervix and 3. patients who had received treatment for the purpose of cure and had not developed a malignant tumor with a known active disease in the previous 5 years);
6. Patients who had received other antitumor therapy (including corticosteroid therapy, immunotherapy) or participated in other clinical studies within 4 weeks before the start of the enrollment (if patients received small-molecule targeted drug therapy, they could be included in the study if the drug was discontinued for more than 5 half-lives), or had not recovered from the previous toxicity;
7. Patients with significant coagulation abnormality;
8. Patients with autoimmune diseases requiring treatment or with a history of syndrome requiring systemic use of steroid immunosuppressive agents, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism, hypothyroidism, etc;
9. Other serious, uncontrolled concomitant diseases that may affect protocol compliance or interfere with results interpretation, including uncontrolled diabetes, or pulmonary disease (a history of interstitial pneumonia, obstructive pulmonary disease, and symptomatic bronchospasm);
10. Evidence of central nervous system disease;
11. Patients who received the live vaccine within 4 weeks of the start of the enrollment;
12. Patients with hepatitis B (HBV HBsAg positive and HBV-DNA≥105), hepatitis C (HCV) infection (HCV antibody positive and HCV-RNA detectable); And subjects with other acquired or congenital immune deficiency diseases, including but not limited to hiv-infected;
13. Pregnant or lactating women;
14. Patients who have had previous organ transplants (except autologous hematopoietic stem cell transplants);
15. Severe or uncontrolled infections;
16. Patients with history of severe neurological or psychiatric illness, including dementia or epilepsy;
17. Patients with drug abuse, medical, psychological or social conditions that may interfere with the study results or the assessment of the study results;
18. Patients are unsuitable for the enrollment according to investigator's judgement.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to two years after the start of the study
  Time from the data of enrollment to of disease progression, or death of any cause, or date of lost follow-up, whichever comes first, otherwise subject data were censored at time last known disease free.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to two years after the start of the study
  Time from the date of enrollment to data of death from any cause, or date of lost follow-up, whichever comes first, and otherwise censored at time last known alive.
incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Since the signing of informed consent forms to 30 days after the last cycle of treatment and 90 days after last dose of anti-PD-1 antibody
  All the adverse events of the patients related will be assessed and graded by NCI CTCAE v 5.0]

OTHER OUTCOMES:
biomarker | the collection of the samples will begin from the signing of informed consent forms（ICF）, and the detection will be competed within 3 months after the last patient discontinued the treatment
  PD-L1, HDAC 3/4/10 expression, circulation tumor DNA（ctDNA）

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Ji, doctor, Principal Investigator — Fudan University; Junning Cao, Doctor, Principal Investigator — Fudan University
Locations (1):
- Dongmei Ji, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No